CLINICAL TRIAL: NCT00428558
Title: A Phase 3 Trial of Systematic Versus Response-adapted Timed-Sequential Induction in Patients With Core Binding Factor (CBF) Acute Myeloid Leukemia (AML)
Brief Title: Timed-Sequential Induction in CBF-AML
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Acute Leukemia French Association (Other); French Innovative Leukemia Organisation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P060504
Record Dates: First submitted 2007-01-29; First posted 2007-01-30 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2007-07

CONDITIONS: Acute Myeloid Leukemia
Keywords: acute myeloid leukemia; Core Binding Factor; t(8;21); inv(16); timed-sequential induction
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Active Comparator): A Phase 3 Trial of Systematic versus Response-adapted Timed-SEQUENTIAL Induction in Patients with Core Binding Factor (CBF) Acute Myeloid Leukemia (AML)
  Interventions: Drug: Chemotherapy (DAUNORUBICINE-CYTARABINE)
- 1 (Experimental): BRAS INDUCTION SEQUENTIAL
  Interventions: Drug: Chemotherapy (DAUNORUBICINE-CYTARABINE)

INTERVENTIONS:
Drug: Chemotherapy (DAUNORUBICINE-CYTARABINE) — A Phase 3 Trial of Systematic versus Response-adapted Timed-SEQUENTIAL Induction in Patients with Core Binding Factor (CBF) Acute Myeloid Leukemia (AML)
  Arms: 2
Drug: Chemotherapy (DAUNORUBICINE-CYTARABINE) — Chemotherapy induction sequential
  Other Names: Chemotherapy induction SEQUENTIAL
  Arms: 1

SUMMARY:
Core binding factor (CBF) acute myeloid leukemias (AML) include AMLs carrying the t(8;21) translocation as well as AMLs carrying either the inversion of chromosome 16 or translocation t(16;16). CBF-AMLs are characterized by their high sensitivity to standard chemotherapeutical agents, especially to cytarabine when administered as high-dose bolus infusions, and thus by a relative good prognosis. However, relapse rates are still comprised between 30 and 50% in these patients, even if overall survival may reach approximately 65% due to the potential salvage of late relapses.

The primary purpose of the protocol is to compare two modalities of timed-sequential induction in order to improve the results of the treatment of CBF-AML patients. This protocol also includes the biological characterization of the heterogeneity of these diseases (gene mutation and transcription profiles), as well as a centralized minimal residual disease monitoring and centralized evaluation of pharmacogenetic polymorphisms.

DETAILED DESCRIPTION:
Core binding factor (CBF) acute myeloid leukemias (AML) include AMLs carrying the t(8;21) translocation as well as AMLs carrying either the inversion of chromosome 16 or translocation t(16;16). CBF-AMLs are characterized by their high sensitivity to standard chemotherapeutical agents, especially to cytarabine when administered as high-dose bolus infusions, and thus by a relative good prognosis. However, relapse rates are still comprised between 30 and 50% in these patients, even if overall survival may reach approximately 65% due to the potential salvage of late relapses. Initial high white blood cell count, activating mutations of cKit, Ras, and FLT3 genes, and persistence of high minimal residual disease (MRD) levels (as evidenced by AML1-ETO or CBFb-MYH11 specific RQ-PCR tools) are the main bad-prognostic factors in patients with CBF-AML.

This project includes a new single French protocol to treat patients with CBF-AML who represent approximately 15% of all AML patients. This common protocol has been elaborated by the two main French cooperative groups for adult AML (ALFA and GOELAMS). In addition to a unique specific therapeutical strategy, this protocol includes the biological characterization of the heterogeneity of these diseases (gene mutation and transcription profiles), as well as a centralized MRD monitoring and centralized evaluation of pharmacogenetic polymorphisms. This project which is well-positioned in the international competition, will use many platforms of the POLECANCER with the following objectives : 1) to improve the results of the treatment of CBF-AML patients; 2) to organize a French clinical and biological network on CBF-AML with the aim to test new targeted therapeutical agents (tyrosine kinase and/or farnesyl transferase inhibitors) in the next future.

TREATMENT DESIGN Induction course Systematic timed-sequential induction (arm A) DAUNORUBICINE (DNR): 60 mg/m2/day IV (30 min), Day 1, 2, and 3 CYTARABINE (AraC): 500 mg/m2/day Continuous infusion, Day 1 to 3 DAUNORUBICINE (DNR): 35 mg/m2/day IV (30 min), Day 8 and 9 CYTARABINE (AraC): 1 gr/m2/12 h IV (2h), Day 8, 9, and 10 Response-adapted timed-sequential induction (arm G) DAUNORUBICINE (DNR): 60 mg/m2/dayIV (30 min), Day 1, 2, and 3 CYTARABINE (AraC): 200 mg/m2/dayContinuous infusion, Day 1 to 7

Peripheral blood and bone marrow evaluation at Day 15. The following second induction course will be administered in patients with persistent marrow disease at Day 15 :

DAUNORUBICINE (DNR): 35 mg/m2/day IV (30 min), Day 16 and 17 CYTARABINE (AraC)1 gr/m2/12 h IV (2h), Day 16, 17, and 18 Persistent marrow disease at Day 15 is defined by more than 10% leukemic blasts in a non aplastic or non very hypoplastic bone marrow aspiration sample.

Salvage course In patients not reaching CR after the first induction course (either SI or TSI), a salvage course will be administered. Salvage therapy should not be initiated before Day 35 of arm A and Day 42 of arm G.

CYTARABINE (AraC) :3 gr/m2/12h IV (2h), Day 1, 3, 5, and 7 AMSACRINE : 100 mg/m2/day IV (30 min), Day 5 to 7 G-CSF lenograstim : from Day 8 until myeloid recovery (> 500 PMN/µL)

Consolidation cycles Three monthly cycles of consolidation will be administered in all patients reaching hematological CR after induction or induction + salvage.

CYTARABINE (AraC): 3 g/m2/12h IV (2h), Day 1, 3, and 5 G-CSF lenograstim : from Day 8 until myeloid recovery (> 500 PMN/µL)

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-60 years.
* With a newly-diagnosed de novo or therapy-related CBF-AML defined

Exclusion Criteria:

* No previously treated with any anti-leukemic agent.
* No presenting any diagnosis of uncontrolled or metastatic tumor.
* OMS performance status < 2,
* Absence of uncontrolled severe infection,
* AST and ALT 2.5 x ULN,
* Total bilirubin 1.5 x ULN,
* Serum creatinine 1.5 x ULN

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2007-07; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study is to increase the Event-free Survival (EFS) | during the 60 months

SECONDARY OUTCOMES:
The complete remission (CR) rate, molecular response (MRD), cumulative incidence of relapse (CIR), disease-free survival (DFS), and overall survival (OS) in both randomization groups. | during the 60 months
The toxicity of both induction strategies (induction deaths and further deaths in first CR). | during the 60 months
The relative prognostic value of : 1) WBC; 2) Mutational status (FLT3, c-Kit, and Ras mutations); and 3) MRD in patient outcome (CR rate, CIR, EFS, DFS, OS). | during the 60 months
The prognostic value of CBF-AML subsets defined on Gene Expression Profiling (GEP) basis. | during the 60 months
The prognostic impact of known polymorphisms of genes involved in the metabolism of cytarabine and anthracyclines (Pharmacogenetic study). | during the 60 months
of patients with CBF-AML through the administration of a systematic | during the 60 months
timed-sequential induction (arm A) as compared to a response-adapted | during the 60 months
timed-sequential induction (arm G). | during the 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Eric JOURDAN, MD,PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Service Hematologie Oncologie, Nîmes, France

REFERENCES:
- [Result] Appelbaum FR, Kopecky KJ, Tallman MS, Slovak ML, Gundacker HM, Kim HT, Dewald GW, Kantarjian HM, Pierce SR, Estey EH. The clinical spectrum of adult acute myeloid leukaemia associated with core binding factor translocations. Br J Haematol. 2006 Oct;135(2):165-73. doi: 10.1111/j.1365-2141.2006.06276.x. Epub 2006 Aug 25. PMID 16939487
- [Derived] Willekens C, Blanchet O, Renneville A, Cornillet-Lefebvre P, Pautas C, Guieze R, Ifrah N, Dombret H, Jourdan E, Preudhomme C, Boissel N; French AML Intergroup. Prospective long-term minimal residual disease monitoring using RQ-PCR in RUNX1-RUNX1T1-positive acute myeloid leukemia: results of the French CBF-2006 trial. Haematologica. 2016 Mar;101(3):328-35. doi: 10.3324/haematol.2015.131946. Epub 2015 Dec 3. PMID 26635039
- [Derived] Duployez N, Nibourel O, Marceau-Renaut A, Willekens C, Helevaut N, Caillault A, Villenet C, Celli-Lebras K, Boissel N, Jourdan E, Dombret H, Figeac M, Preudhomme C, Renneville A. Minimal residual disease monitoring in t(8;21) acute myeloid leukemia based on RUNX1-RUNX1T1 fusion quantification on genomic DNA. Am J Hematol. 2014 Jun;89(6):610-5. doi: 10.1002/ajh.23696. Epub 2014 Mar 8. PMID 24616160
- [Derived] Jourdan E, Boissel N, Chevret S, Delabesse E, Renneville A, Cornillet P, Blanchet O, Cayuela JM, Recher C, Raffoux E, Delaunay J, Pigneux A, Bulabois CE, Berthon C, Pautas C, Vey N, Lioure B, Thomas X, Luquet I, Terre C, Guardiola P, Bene MC, Preudhomme C, Ifrah N, Dombret H; French AML Intergroup. Prospective evaluation of gene mutations and minimal residual disease in patients with core binding factor acute myeloid leukemia. Blood. 2013 Mar 21;121(12):2213-23. doi: 10.1182/blood-2012-10-462879. Epub 2013 Jan 15. PMID 23321257